CLINICAL TRIAL: NCT04838106
Title: Outcomes of Patients Who Survived Treatment on an Intensive Care Unit for COVID-19 in England and Wales: a Comparative Retrospective Cohort Study (OPTIC-19)
Brief Title: Outcomes of Patients Who Survived Treatment on an Intensive Care Unit for COVID-19 in England and Wales
Acronym: OPTIC-19
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Intensive Care National Audit & Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: PID15456; 21/SC/0021 (Other: South Central - Hampshire B Research Ethics Committee); 21/CAG/0017 (Other: Confidentiality Advisory Group)
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Covid19; Myocardial Infarction; Stroke; Critical Illness; Heart Failure; Deep Vein Thrombosis; Pulmonary Embolism; Renal Failure
MeSH Terms: conditions — COVID-19; Myocardial Infarction; Stroke; Critical Illness; Heart Failure; Venous Thrombosis; Pulmonary Embolism; Renal Insufficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid19: Patients admitted to an adult (16 years or over), general ICU in England or Wales as an emergency with confirmed COVID-19 between 1st January to 1st July 2020.
  Interventions: Other: Not applicable as observational study
- Non Covid19: Patients admitted to an adult (16 years or over), general ICU in England or Wales as an emergency without confirmed COVID-19 between 1st July 2016 and 1st July 2020.
  Interventions: Other: Not applicable as observational study

INTERVENTIONS:
Other: Not applicable as observational study — Not applicable as observational study.

SUMMARY:
This retrospective cohort study aims to characterise outcomes for patients treated on an intensive care unit (ICU) with COVID-19 in England and Wales, one year after discharge from hospital. Outcomes will be compared with patients admitted as an emergency to an ICU for other conditions. The study will use existing national audit data linked to routine healthcare datasets.

DETAILED DESCRIPTION:
Across England and Wales, over 10,000 patients have been treated for severe coronavirus disease 2019 (COVID-19) on an intensive care unit. Around 60% survived to leave hospital. It is unknown how survivors' severe COVID-19 infection, or the treatment they received on the intensive care unit, will affect their long-term health. Understanding what happens to these patients can help ensure they receive suitable care from their General Practitioner (GP) and other National Health Service (NHS) services after they leave hospital.

This study will follow up survivors for 1 year after discharge from hospital. The investigators will use data collected by the Intensive Care National Audit and Research Centre (ICNARC) to identify patients who were treated on an ICU for COVID-19. The investigators will then use NHS data to see whether these patients were readmitted to hospital and why. Information from the Office of National Statistics will identify whether patients died. By linking different sources of patient data, the investigators will estimate the health risks faced by survivors of severe COVID-19. These risks will be compared to those in patients treated on an ICU for other conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or over
* Admitted to an adult, general ICU in England or Wales as an emergency (unplanned)
* Admitted to ICU for either: a) confirmed COVID-19 between 1st January to 1st July 2020 or b) without confirmed COVID-19 between 1st July 2016 and 1st July 2020-

Exclusion Criteria:

* Patients who died in hospital after treatment on an ICU

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to an adult (16 years or over), general ICU in England or Wales as an emergency between 1st July 2016 and 1st July 2020 who survived to hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 319600 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | One year
  Mortality after discharge from hospital

SECONDARY OUTCOMES:
Rate of emergency hospital admission | one year
  Emergency hospital admission
Rate of emergency hospital admission for respiratory infection | one year
  Emergency hospital admission for respiratory infection
Rate of emergency hospital admission for a major adverse cardiac event | one year
  Emergency hospital admission for a major adverse cardiac event (myocardial infarction, stroke, heart failure)
Rate of emergency hospital admission for a venous thrombotic event | one year
  Emergency hospital admission for a venous thrombotic event (deep vein thrombosis or pulmonary embolism)
Rate of development of end stage renal failure | one year
  Development of end stage renal failure treated by renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Watkinson, MD, Principal Investigator — University of Oxford
Locations (1):
- Critical Care Research Group, Nuffield Department of Clinical Neurosciences, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available due to privacy and legal implications.

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04838106/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04838106/SAP_001.pdf